CLINICAL TRIAL: NCT02438644
Title: Observational Study of the Effectiveness and Safety of Vismodegib (Erivedge) in Patients Treated in Argentina
Brief Title: Observational Study of Vismodegib (Erivedge) in Patients Treated in Argentina
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29740
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study Population: Patients who are prescribed vismodegib in Argentina, according to standard of care and in line with the current SPC and local labeling, are eligible for observation. Dosing and treatment duration of vismodegib are at the discretion of the physician in accordance with local clinical practice and local labeling. Only patients with laBCC or mBCC will be considered in the effectiveness analysis.

SUMMARY:
This observational, noninterventional study is designed to further characterize the effectiveness and safety profile of vismodegib (Erivedge) in Argentine patients. Only patients with locally advanced basal cell carcinoma (laBCC) or metastatic basal cell carcinoma (mBCC) will be considered in the effectiveness analysis. Study duration is estimated to be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Argetine patients prescribed vismodegib according to standard of care and in line with Summary of Product Characteristics (SPC) and local labeling
* Diagnosis of laBCC or mBCC for the effectiveness analysis

Exclusion Criteria:

* None specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is characterized by patients who are prescribed vismodegib in Argentina, according to standard of care and in line with the current SPC and local labeling. Data collection will be prospective except in the cases when a treating physician contacts the vendor for the first time after the patient has started treatment with vismodegib. In these cases the vendor will retrospectively collect data from the start of treatment. Only patients with laBCC or mBCC will be considered in the effectiveness analysis.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Response rate as assessed by the treating physician | Approximately 12 months

SECONDARY OUTCOMES:
Duration of treatment | Approximately 12 months
Duration of response as assessed by the treating physician | Approximately 12 months
Incidence of adverse events | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Undecided